CLINICAL TRIAL: NCT00308633
Title: Mechanism and Vascular Effects of Endothelial Progenitor Cell Mobilization in Patients With Coronary Artery Disease Undergoing Cardiac Rehabilitation
Brief Title: Endothelial Progenitor Cells and Nitric Oxide in Cardiac Rehabilitation Program Participants
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060122; 06-H-0122
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-30

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Cardiac Rehabilitation; Apoptosis; Gene Expression; Nitric Oxide; Reactive Oxygen Species; Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease

SUMMARY:
This study will measure blood levels of endothelial progenitor cells (EPCs) and nitric oxide (NO) in patients with coronary artery disease (CAD) who are participating in a 3-month cardiac rehabilitation program at Suburban Hospital in Bethesda, MD. EPCs are a kind of stem cell produced by the bone marrow that can develop into cells found in arteries and in the heart and, therefore, can repair diseased vessels. The study will examine whether the EPCs are affected by exercise and will look at how they may contribute to repair of cells lining the diseased arteries as a result of participation in the rehabilitation program.

People with coronary artery disease may be eligible for this study. Candidates are screened with a medical history, physical examination, electrocardiogram, and blood tests. CAD patients also to a treadmill exercise test.

Volunteers' participation ends at the screening visit. The blood drawn at screening is used to identify EPC specific genes to compare with the EPC genes from patients with CAD.

CAD patients participate in Suburban Hospital's cardiac rehabilitation program. The exercise portion of the program includes 36 sessions of about 60 minutes each, spaced over approximately 3 months. Patients have a baseline blood test at screening and repeat blood tests at the end of each month of participation in the rehabilitation program. Some of the blood will be used for genetic tests to see how genes of the EPCs are changed by the patient's participation in the rehabilitation program.

DETAILED DESCRIPTION:
Exercise training has long been recommended as a means of improving effort tolerance and reducing morbidity and mortality in patients with coronary artery disease (CAD). One mechanism of benefit may be through improved endothelial function with enhanced nitric oxide (NO) bioactivity. Such an effect may augment blood flow to exercising skeletal muscle and to the myocardium, and reduce vascular inflammation, platelet activation and adherence which could diminish the risk of thrombosis. In 46 patients with CAD, participating in the Suburban Hospital cardiac rehabilitation program (Protocol 03-H-0086), we detected increases in circulating endothelial progenitor cells (EPCs), which may have the capacity to repair diseased or dysfunctional endothelium. In the last 23 participants (following amendment of the protocol) a subset showed increase in whole blood nitrite - a marker of intravascular NO - at completion of program. However, not all patients showed EPC mobilization or increased intravascular NO despite compliant program participation and improved effort tolerance. One possibility is that EPCs from patients who fail to derive vascular benefit as evidenced by increased intravascular NO may have different EPC gene expression profiles at baseline or in response to repetitive exercise, resulting in diminished protection of EPCs against oxidant stress with initiation of apoptosis, compared with EPC gene expression in patients who show evidence of EPC mobilization and endothelial repair. The purpose of our study is to 1) Prospectively demonstrate a relationship between EPC mobilization and increased whole blood nitrite as a marker of improved vascular NO bioactivity due to EPC mobilization, and 2) Determine EPC gene expression profiles, with a focus on activation or suppression of genes whose products regulate intravascular redox potential, apoptosis and growth factor and cytokine secretion. We hypothesize that activation or suppression of critical genes in EPCs at baseline or during exercise may determine EPC mobilization, endothelial differentiation and vascular repair potential as evidenced by increased intravascular NO.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults older than 21 years.

Coronary artery disease established by angiography.

At least two months interval since myocardial infarction or coronary artery bypass surgery.

At least one month interval since percutaneous coronary intervention or congestive heart failure symptoms.

No medical condition that might prohibit safe participation in cardiac rehabilitation.

Subject understands protocol and provides written, informed consent in addition to willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

Significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease) as determined by echocardiography.

Angina pectoris that is prolonged in duration (greater than 20 minutes), or does not respond to nitroglycerin (2 tablets) within 2 weeks of referral to the program.

Subjects physically unable to perform cardiac rehabilitation protocol due to neurologic or orthopedic conditions.

Women of childbearing age unless recent pregnancy test is negative.

Lactating women.

Implantable cardioverter-defibrillator (ICD)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2006-03-23; Primary Completion 2007-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Dimmeler S, Aicher A, Vasa M, Mildner-Rihm C, Adler K, Tiemann M, Rutten H, Fichtlscherer S, Martin H, Zeiher AM. HMG-CoA reductase inhibitors (statins) increase endothelial progenitor cells via the PI 3-kinase/Akt pathway. J Clin Invest. 2001 Aug;108(3):391-7. doi: 10.1172/JCI13152. PMID 11489932
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076